CLINICAL TRIAL: NCT00329355
Title: A Randomized, Double-blind, Single Migraine Attack, Placebo-controlled, Parallel-group Multicenter Study to Evaluate the Efficacy and Tolerability of Trexima (Sumatriptan Succinate.Naproxen Sodium) Tablets vs Placebo When Administered During the Mild Pain Phase of Menstrual Migraine in Women With Dysmenorrhea
Brief Title: Menstrual Migraine Treatment With TREXIMET (Formerly Known as TREXIMA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRX105852
Record Dates: First submitted 2006-05-22; First posted 2006-05-24 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Migraine; Migraine Disorders
Keywords: menstrual migraine; headache; early intervention; dysmenorrhea
MeSH Terms: conditions — Migraine Disorders; Headache; Dysmenorrhea | interventions — Sumatriptan; Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: sumatriptan succinate/naproxen sodium

SUMMARY:
This study was designed to determine efficacy of TREXIMET (sumatriptan/naproxen sodium), formerly known as TREXIMA compared to placebo for the treatment of a menstrual migraine.

DETAILED DESCRIPTION:
A randomized, double-blind, single migraine attack, placebo-controlled, parallel-group, multicenter study to evaluate the efficacy and tolerability of TREXIMA* (sumatriptan succinate/naproxen sodium) tablets vs placebo when administered during the mild pain phase of menstrual migraine in women with dysmenorrhea (*TREXIMET)

ELIGIBILITY:
Inclusion Criteria:

* At least a 6 month history of physician diagnosed migraine and typically experiences 2-6 migraine attacks per month
* Typically experiences moderate to severe migraine pain preceded by a mild pain phase
* Differentiate between mild migraine pain and other headache types
* Women of childbearing potential must be on adequate contraception

Exclusion Criteria:

* Pregnant and/or nursing mother
* History of cardiovascular disease
* Uncontrolled hypertension
* Basilar or Hemiplegic migraine
* History of stroke or transient ischemic attacks (TIA)
* History of epilepsy or treated with anti-epileptics within past 5 years
* Impaired hepatic or renal function
* History of gastrointestinal bleeding or ulceration
* Allergy or hypersensitivity to aspirin or any other NSAID
* Allergy or hypersensitivity to triptans
* Participated in an investigational drug trial in the previous 4 weeks

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2006-05; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Score on a 4-pt migraine pain scale for a single menstrual migraine attack | 2 to 48 hours

SECONDARY OUTCOMES:
Freedom from all migraine pain and symptoms, satisfaction, presence or absence of neck pain/discomfort, sinus pain/pressure, menstrual symptoms, recurrence of head pain, safety and tolerability | 2 to 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (33):
- United States (33):
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Irvine, California
  - GSK Investigational Site, Redondo Beach, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Boulder, Colorado
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Port Orange, Florida
  - GSK Investigational Site, Sunrise, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, West Chester, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Carnegie, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Warwick, Rhode Island
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Georgetown, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Result] Durham PL, Vause CV, Derosier F, McDonald S, Cady R, Martin V. Changes in salivary prostaglandin levels during menstrual migraine with associated dysmenorrhea. Headache. 2010 May;50(5):844-51. doi: 10.1111/j.1526-4610.2010.01657.x. Epub 2010 Mar 26. PMID 20353434
- [Result] Mannix LK, Martin VT, Cady RK, Diamond ML, Lener SE, White JD, Derosier FJ, McDonald SA. Combination treatment for menstrual migraine and dysmenorrhea using sumatriptan-naproxen: two randomized controlled trials. Obstet Gynecol. 2009 Jul;114(1):106-113. doi: 10.1097/AOG.0b013e3181a98e4d. PMID 19546766
- [Derived] Martin VT, Ballard J, Diamond MP, Mannix LK, Derosier FJ, Lener SE, Krishen A, McDonald SA. Relief of menstrual symptoms and migraine with a single-tablet formulation of sumatriptan and naproxen sodium. J Womens Health (Larchmt). 2014 May;23(5):389-96. doi: 10.1089/jwh.2013.4577. Epub 2014 Feb 28. PMID 24579886
- [Derived] Cady RK, Diamond ML, Diamond MP, Ballard JE, Lener ME, Dorner DP, Derosier FJ, McDonald SA, White J, Runken MC. Sumatriptan-naproxen sodium for menstrual migraine and dysmenorrhea: satisfaction, productivity, and functional disability outcomes. Headache. 2011 May;51(5):664-73. doi: 10.1111/j.1526-4610.2011.01894.x. PMID 21521204
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: TRX105852 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: TRX105852 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: TRX105852 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: TRX105852 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: TRX105852 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: TRX105852 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: TRX105852 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register